CLINICAL TRIAL: NCT06627322
Title: Registry Based Randomized Controlled Trial of Multiple Combination Strategies of Intensive Glycemic Control to Reduce a Composite of Macrovascular and Microvascular Events in Type 2 Diabetes With Cardiovascular Risk Factors (REMATCH Study)
Brief Title: A Registry-based Randomized Controlled Trial in Type 2 Diabetes With Cardiovascular Risk Factors (REMATCH)
Acronym: REMATCH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kyu Chang Won (Other)
Collaborators: Boryung Pharmaceutical Co., Ltd (Industry); Dong-A ST Co., Ltd. (Industry); HK inno.N Corporation (Industry); Daewoong Pharmaceutical Co. LTD. (Industry); Chong Kun Dang Pharmaceutical Corp. (Industry); Celltrion (Industry); Kakao Healthcare Corp. (Unknown); Handok Inc. (Industry)
Responsible Party: Sponsor-Investigator, Kyu Chang Won, Professor, Yeungnam University Hospital
Organization: Yeungnam University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: YUMC 2023-08-009
Record Dates: First submitted 2024-09-26; First posted 2024-10-04 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; T2D; T2DM; RRCT
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: RRCT (Registry-based randomized controlled trial)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard treatment arm (HbA1c 7.0% target) (Active Comparator): Metformin/DPP-4i-based or Metformin/SGLT2i-based dual-combination therapy. Treatment and Follow-up : Maximum 4 years
  Interventions: Drug: Dual-combination therapy
- Intensive treatment arm (HbA1c 6.0% target): plus real-time CGM (Experimental): Randomly assigned into 2 sub-groups Device: Dexcom G7 plus Kakaohealthcare Pasta. (Barozen Fit is also available.) Treatment and Follow-up : Maximum 4 years
  Interventions: Drug: Triple-combination therapy; Device: Dexcom G7, Pasta

INTERVENTIONS:
Drug: Dual-combination therapy — Group 1: Metformin/DPP-4i-based or Metformin/SGLT2i-based dual-combination therapy. Any oral antiglycemic drugs on the market.
  Arms: Standard treatment arm (HbA1c 7.0% target)
Drug: Triple-combination therapy — Group 2: Metformin/SGLT2i/DPP-4i-based triple-cobmination therapy, or Group 3: Metformin/SGLT2i/Thiazolidinedione-based triple-cobmination therapy Any oral antiglycemic drugs on the market.
  Arms: Intensive treatment arm (HbA1c 6.0% target): plus real-time CGM
Device: Dexcom G7, Pasta — Real-time continous glucose monitoring system (CGMS) Device (sensor): Dexcom G7 Device (software): Kakaohealthcare Pasta Barozen Fit is also available.
  Arms: Intensive treatment arm (HbA1c 6.0% target): plus real-time CGM

SUMMARY:
Glycemic control is a mainstay of diabetes management to reduce the risk of microvascular complications and cardiovascular outcomes in people with type 2 diabetes (T2D). However, intensive control to near-normal glycated hemoglobin (HbA1c) yielded complex results in previous landmark trials. Potential risks of intensive glycemic control, such as hypoglycemia and weight gain, may partly contributed to the possible harms associated with this approach. Recent advances in diabetes management with development of newer antidiabetic drugs which minimize possible harms of intensive glycemic control as well as reduce cardiorenal risks enabled safer glycemic reduction. Thus, this randomized trial aims to evaluate the effects of near normalization of HbA1c with novel approaches on microvascular complications and cardiovascular outcomes in people with T2D.

DETAILED DESCRIPTION:
This is a multicenter, prospective, registry-based, randomized, open-label, active-comparator controlled trial involving 5,950 eligible participants with T2D, cardiovascular risk factors, and elevated HbA1c (≥7.0%). Participants will be randomly assigned to either intensive arm (targeting 6.0% of HbA1c) or standard arm (targeting 7.0% of HbA1c). The primary end point is the time to development of a composite of major adverse cardiovascular and diabetic microvascular events.

This study is designed as registry-based randomized clinical trial (RRCT), which adheres to the characteristics of both randomized clinical trial and registry-based prospective observational study. The participants will be randomly assigned into either intensive glycemic control arm or standard glycemic control arm, and the outcomes and variables will be recorded by multiple registries including hospital electronic medical records, nationwide health registry (the national health insurance service, NHIS), and Korean Statistical Information Service registry.

ELIGIBILITY:
Inclusion Criteria:

1. ≥19 years of age
2. Patient agreed to participate in the study and signed a written informed consent form
3. Type 2 diabetes (ADA criteria)
4. HbA1c≥7.0% and <10.0% in patients receiving monotherapy, dual-combination therapy, or triple-combination therapy (when the submaximal dose was administered) with oral antidiabetic drugs (OADs)
5. Any of the following:

A. Patients who one or more of the following conditions

1. Coronary artery disease
2. Atherosclerotic ischemic stroke, transient ischemic attack, carotid artery disease, peripheral artery disease, abdominal aortic aneurysm
3. Prevalence of diabetes ≥10 years
4. Left ventricular hypertrophy
5. Albuminuria
6. Chronic kidney disease (eGFR<60mL/min/1.73m²)
7. Diabetic Retinopathy
8. Diabetic neuropathy or B. Patients who have two or more of the following cardiovascular risk factors

(1) Family history of early-onset ASCVD (first-degree relatives with disease before age 55 for men and before age 65 for women) (2) Hypertension (on medication or with SBP≥140 mm Hg or DBP≥90 mm Hg) (3) Low HDL cholesterol concentration (<40 mg/dL) (4) Current smoker (5) Obese (BMI≥25 kg/m²)

Exclusion Criteria:

1. Type 1 diabetes
2. Estimated GFR<45 ml/min/1.73m²
3. AST or ALT greater than 3 times the normal upper limit
4. Symptomatic heart failure (NYHA Class III or IV)
5. History of hospitalization for acute cardiovascular events within 3 months prior to the date of consent
6. Currently in active treatment for malignancy
7. Contraindications for each assigned drug, as applicable
8. Pregnant and nursing women
9. If the investigator determines that assignment to the standard glycemic control arm raises ethical concerns

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5950 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
A composite of major adverse cardiovascular events (MACE) or diabetic microvascular events | 6-month, 1-, 2-, 3-, 4-year after enrollment
  The time from the date of randomization to the first occurrence of any of the events or records in A** and B** as defined below.
  [**A.Major adverse cardiovascular events (MACEs): (1) Death from cardiovascular causes (2) Non-fatal stroke (3) Non-fatal myocardial infarction (4) Hospitalization due to unstable angina (5) Hospitalization due to heart failure (6) Hospitalization due to peripheral artery disease (7) Coronary or peripheral revascularization
  **B.Diabetic microvascular events
  * B1. A composite of kidney events:
    1. Death from kidney causes
    2. Development of end-stage renal disease
    3. Sustained decline in eGFR of 40% or more from baseline
    4. Occurrence of marked albuminuria,
  * B2. A composite of eye events:
    1. Development or progression of diabetic retinopathy (proliferative diabetic retinopathy or macular edema)
    2. Blindness due to diabetic retinopathy
    3. Surgical treatment of diabetic retinopathy or intravitreal injections]

SECONDARY OUTCOMES:
Composite endpoint of cardiorenal events_#1 | 6-month, 1-, 2-, 3-, 4-year after enrollment
  Time from the date of randomization to the first occurrence of any of the events or histories of A** or B** defined in the protocol. [**A. Major cardiovascular events : (1) Death from cardiovascular cause, (2) Non-fatal stroke, (3) Non-fatal myocardial infarction, (4) hospitalization due to heart failure; **B. Major Kidney Events: (1) Death from kidney causes, (2) Development of end-stage renal disease, (3) Sustained decline in eGFR of 40% or more from baseline]
Composite endpoint of cardiorenal events_#2 | 6-month, 1-, 2-, 3-, 4-year after enrollment
  Time from the date of randomization to the first occurrence of any of the events or histories of A [is equal to the "A" defined in the primary endpoint] or B [is equal to the "B1" defined in the primary endpoint] defined in the protocol.
Level of HbA1c (glycated haemoglobin) | 6-month, 1-, 2-, 3-, 4-year after enrollment
  The level is a crucial indicator for managing Type 2 Diabetes. It is used to assess long-term blood sugar control and the effectiveness of your diabetes management strategies.
The proportion of participants who exhibited a weight change (either gain or loss) of 10% or more | 6-month, 1-, 2-, 3-, 4-year after enrollment
Change in waist circumference at each time point from baseline | 6-month, 1-, 2-, 3-, 4-year after enrollment
  Abdominal obesity is assessed by measuring waist circumference. Long-term follow-up studies have reported that abdominal obesity increases the risk of type 2 diabetes, cardiovascular disease, and death, even after correction for body mass index (BMI).
Change in estimated glomerular filtration rate (eGFR) from baseline | 6-month, 1-, 2-, 3-, 4-year after enrollment
  Glomerular filtration rate (GFR) is a measure of how well your kidneys are functioning. It estimates the amount of blood that pass through the glomeruli (the tiny filters in the kidneys) each minute. Estimated GFR will be calcuated by CKD-EPI formula in this study.
Change in lipid panel | 6-month, 1-, 2-, 3-, 4-year after enrollment
  Lipid panel: blood total cholesterol, LDL-cholesterol, HDL-cholesterol, Tryglycerides.
Change in urine albumin to creatinine ratio (UACR) from baseline | 6-month, 1-, 2-, 3-, 4-year after enrollment
  The urine albumin to creatinine ration (UACR) is a test that measures the amount of albumin (a typie of protein) in the urine relative to the amount of creatinine. It is used to assess your kidney function, particularly to detect early signs of kidney damage or disease.
Safety endopoints | 6-month, 1-, 2-, 3-, 4-year after enrollment
  Incidence rate and charateristics (causality, seriousness, severity, outcomes, action taken etc.) of adverse events, serious adverse events, and adverse events of special interest (acute kidney injury, hypoglycemia, acute hyperglycemic complications, GI symptoms, ,urogenital infection, edema, weight gain)

CONTACTS AND LOCATIONS:
Overall Officials: Kyu Chang Won, M.D., Ph.D., Principal Investigator — Yeungnam University Hospital
Locations (2):
- South Korea (2):
  - Yeungnam University Medical Center, Daegu
  - Korea University Anam Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No